CLINICAL TRIAL: NCT03304821
Title: Granulocyte-Macrophage Stimulating Factor (GM-CSF) in Peripheral Arterial Disease: The GPAD-3 Study
Brief Title: Granulocyte-Macrophage Stimulating Factor (GM-CSF) in Peripheral Arterial Disease
Acronym: GPAD-3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00087198; 1R61HL138657 (NIH)
Record Dates: First submitted 2017-10-04; First posted 2017-10-09 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Peripheral Artery Disease (PAD)
Keywords: Atherosclerotic peripheral artery disease; Granulocyte-macrophage colony stimulating factor (GM-CSF); Atherosclerosis; Cardiology; Vascular disease
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis; Vascular Diseases | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Intervention Model Description: Participants will be randomized, in a 2:1 manner, to receive:
  * Group A: Subcutaneous GM-CSF 500µg on Monday, Wednesday, Friday (n=117)
  * Group B: Placebo on Monday, Wednesday, Friday (n=59)
  Participants will be stratified on diabetes status ensuring that a proportionate number of diabetics (2:1) are randomized to each group.
Who Masked: Participant, Investigator
Masking Description: Participants and the primary investigator will be blinded to group assignment. Blinding will be maintained by Investigational Pharmacy and blood counts will be reviewed by one of the study co-investigators who will make dose-modifications, when necessary.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GM-CSF (Experimental): Participants receiving 500µg of granulocyte-macrophage colony stimulating factor (GM-CSF), administered subcutaneously. Prior to randomization to a study arm, eligible participants will be trained to perform subcutaneous injections and instructed to walk at least three times a day until they develop claudication or symptomatic limitation for 4 weeks.
  Interventions: Drug: GM-CSF
- Placebo (Placebo Comparator): Participants receiving 500µg of a placebo, administered subcutaneously. Prior to randomization to a study arm, eligible participants will be trained to perform subcutaneous injections and instructed to walk at least three times a day until they develop claudication or symptomatic limitation for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GM-CSF — Participants will self-administer 500 μg/day of GM-CSF, subcutaneously, three times per week (Monday, Wednesday, Friday) for three weeks. After three months the participants will receive a second administration of 500 μg/day of subcutaneous GM-CSF, three times per week for another 3 weeks and then will be followed for another 3 months.
  Other Names: Sargramostim; Leukine
  Arms: GM-CSF
Drug: Placebo — Participants will self-administer 500 μg/day of a placebo, subcutaneously, three times per week (Monday, Wednesday, Friday) for three weeks. After three months the participants will receive a second administration of 500 μg/day of a placebo administered subcutaneously, three times per week for another 3 weeks and then will be followed for another 3 months.
  Arms: Placebo

SUMMARY:
Peripheral artery disease (PAD) is a disease in which plaque builds up in the arteries that carry blood to the head, organs, and limbs. PAD usually occurs in the arteries in the legs, but can affect any arteries. Over time, plaque can harden and narrow the arteries which limits the flow of oxygen-rich blood to organs and other parts of the body. Blocked blood flow to the arteries can cause pain and numbness. The pain is usually worse with exercise and gets better with rest. PAD can raise the risk of getting an infection which could lead to tissue death and amputation. This study is investigating whether granulocyte-macrophage colony stimulating factor (GM-CSF) improves symptoms and blood flow in people with PAD. GM-CSF is a drug that is used to stimulate the bone marrow to release stem cells. Participants in the study will be randomly selected to receive GM-CSF or a placebo. After a four-week screening phase, participants will receive injections of GM-CSF or a placebo three times a week for three-weeks. Three months later, participants will again receive injections of GM-CSF or placebo three times a week for three-weeks. At six months, the study team will follow up to see if the group that received GM-CSF had more improvement than the group that received placebo.

DETAILED DESCRIPTION:
Atherosclerotic peripheral artery disease (PAD) of the lower extremities afflicts up to 8% of the U.S. population and lack of adequate sustainable therapies necessarily results in severe morbidity and increased mortality. Both experimental and current clinical data indicate that GM-CSF has the capacity to mobilize a variety of progenitor cells (PCs), including endothelial PCs that appear to improve ischemia.

This study builds on the findings of prior research which showed improvements in claudication symptoms after treatment with GM-CSF. This study aims to answer whether repeat administration of GM-CSF at 3 months will further improve symptoms. The researchers will investigate in a double-blind placebo-controlled randomized study whether 3 weeks of three-times-a-week injection of GM-CSF will improve measures of ischemia in patients with intermittent claudication.

This study will recruit 176 participants with atherosclerotic PAD and claudication. After screening for inclusion and exclusion criteria, eligible subjects will be trained to perform subcutaneous injections and instructed to walk until they develop claudication or symptomatic limitation at least three times a day for 4 weeks. At the end of the 4-week period, subjects will undergo baseline testing and will be randomized to receive 500 μg/day of GM-CSF thrice weekly for 3 weeks (group A) or a placebo (group B). After 3 months, follow-up endpoint testing will be performed. Subjects in group A will then receive the second administration of 500 μg/day of subcutaneous GM-CSF thrice weekly for another 3 weeks and be followed for another 3 months for endpoint measurements, while Group B subjects will receive a matching placebo. The primary outcome is change in walking performance in the active treatment group after 6 months compared to the placebo group. The secondary outcome includes change in peak walking time at 6 months, changes in circulating progenitor cell levels, ankle brachial index (ABI), walking impairment questionnaire (WIQ) scores, and 36-item Short-Form Health Survey (SF-36) scores. Long-term follow up, by way of a telephone call, will occur with each participant one, two and three years after they enrolled in the study to administer questionnaires and collect adverse event data.

In response to the Coronavirus Disease 2019 (COVID-19) crisis on April 3, 2020 the Institutional Review Board (IRB) approved temporary modifications to this study to postpone study visits that do not involve active drug/placebo use.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects must be (a) post-menopausal, (b) surgically sterile or (c) use adequate birth control and have a negative pregnancy test within 3 days prior to administration of study drug and should not be breastfeeding.
* Documented symptomatic PAD
* Clinically stable (at least 2 months prior to enrollment) history of intermittent claudication or walking impairment (Rutherford Class II) with no change in symptom severity in the 2 months prior to screening.
* On statin therapy for previous 3 months prior to enrollment, unless statin intolerant.
* Peak Walking Time (PWT) between 1 and 12 minutes on a standardized Gardner treadmill protocol or modified Gardner protocol or less than 12 minutes on a modified Bruce protocol in case PWT on Gardner protocol is more than 12 minutes.
* A Doppler-derived ankle-brachial index (ABI) of < 0.90 in the symptomatic limb after 10 minutes of rest at screening. For subjects with an ABI of >1.3 (non-compressible arteries) a Toe-Brachial Index (TBI) of < 0.70 must be obtained for subject qualification, or if ABI is > 0.9 to 1.0 , and a reduction of 20% in ABI measured within 1 minute of treadmill testing.
* On appropriate and stable medical therapy for atherosclerosis for at least 2 months prior to enrollment.
* Able to give informed consent.
* Diabetics with a dilated eye exam excluding proliferative retinopathy in the previous 12 months prior to enrollment.

Exclusion Criteria:

* Recent or current active infections (treated with antibiotics)
* Recent (6 months prior to randomization) or current active cancer undergoing treatment
* Recent (3 months prior to randomization) change in statin or cilostazol therapy
* Critical limb ischemia either chronic (Rutherford Class >II) or acute ischemia manifested by rest pain, ulceration, or gangrene
* Recent (3 months prior to randomization) lower extremity vascular surgery, angioplasty or lumbar sympathectomy
* Planned participation in a structured exercise treatment protocol in the future or within period of study
* Prior myeloid malignancy
* Recent (3 months prior to randomization) Unstable angina, myocardial infarction, transient ischemic attack (TIA), stroke or revascularization
* Severe heart failure (Class III or IV) or heart muscle disease
* Limitation on exercise for symptoms other than intermittent claudication such as arthritis or dyspnea
* Below- or above-knee amputation; wheelchair confinement
* Use of a walking aid other than a cane
* Walking impairment for reasons other than PAD e.g. Parkinson's disease
* Uncontrolled diabetes mellitus (defined as HbA1c > 10.0)
* Chronic renal disease (creatinine of >2.5 mg/dl) or hepatic disease (> 3 X elevations in aspartate aminotransferase (AST) and alanine aminotransferase (ALT))
* White blood cell count < 3k/cmm
* Hemoglobin (HGB) < 10g/dL
* Blood Pressure Systolic >180 and/or Diastolic >100
* Taking Immunosuppressant drugs
* Ophthalmologic conditions associated with a neo-vascular response
* Alcohol or drug abuse, or any other disease process that, in the opinion of the PI, will interfere with the ability of the patient to participate in the study
* Inability to attend study visits

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2017-12-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in 6-minute walk distance | Baseline, Month 3, Month 6, Month 9
  Participants will be walk up and down a 100-foot hallway for 6 minutes to cover the maximum distance possible. The distance, measured in feet, completed after 6 minutes will be recorded.

SECONDARY OUTCOMES:
Change in Peak Walking Time (PWT) | Baseline, Month 3, Month 6, Month 9
  Graded treadmill exercise testing will be performed using the Gardner protocol where the treadmill speed is kept at 2 mph and the grade starts at 0 and inclines by 2% every two minutes. The peak walking time (PWT) is the time until exercise is terminated because of severe claudication. Exercise testing will be performed twice and longest time will be used as the PWT for that study visit.
Change in Walking Impairment Questionnaire (WIQ): Walking Distance Score | Baseline, Month 3, Month 6, Month 9, Follow-up Years 1, 2, and 3
  The Walking Impairment Questionnaire (WIQ) domain of walking distance asks respondents to rate how difficult it is to walk around home, as well as distances of 50, 150, 300, 600, 900 and 1500 feet. Possible responses are: not hard (4), slightly difficult (3), somewhat difficult (2), very difficult (1), and unable to do (0). Total raw scores range from 0 to 28 with higher scores indicating increased ability to walk further distances.
Change in Walking Impairment Questionnaire (WIQ): Walking Speed Score | Baseline, Month 3, Month 6, Month 9, Follow-up Years 1, 2, and 3
  The Walking Impairment Questionnaire (WIQ) domain of walking speed asks respondents to rate how difficult it is to walk the distance of one block slowly, at an average speed, quickly, and running/jogging. Possible responses are: not hard (4), slightly difficult (3), somewhat difficult (2), very difficult (1), and unable to do (0). Total raw scores range from 0 to 16 with higher scores indicating increased ability to walk fast.
Change in Walking Impairment Questionnaire (WIQ): Stair Climbing Score | Baseline, Month 3, Month 6, Month 9, Follow-up Years 1, 2, and 3
  The Walking Impairment Questionnaire (WIQ) domain of stair climbing asks respondents to rate how difficult it is to climb 1, 2, and 3 flights of stairs. Possible responses are: not hard (4), slightly difficult (3), somewhat difficult (2), very difficult (1), and unable to do (0). Total raw scores range from 0 to 12 with higher scores indicating better ability to climb stairs.
Change in 36-item Short-Form Health Survey (SF-36) Score | Baseline, Month 3, Month 6, Month 9, Follow-up Years 1, 2, and 3
  36-item Short-Form Health Survey (SF-36) consists of eight scaled scores for the domains of: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Study participants respond to questions relating to their health and activity level by selecting from a variety of Likert scale and yes/no response options. Each scale is directly transformed into a 0-100 scale and lower scores indicate more disability (a score of 0 equates to maximum disability while a score of 100 indicates no disability).
Change in Claudication Onset Time (COT) | Baseline, Month 3, Month 6, Month 9
  Claudication onset time (COT) during the treadmill exercise will be recorded along with the peak walking time (PWT). The claudication onset time (COT) is the duration of exercise until onset of the participant's typical claudication. This is differentiated from the peak walking time (PWT) which is the time until exercise is terminated because of severe claudication. Graded treadmill exercise testing will be performed using the Gardner protocol where the treadmill speed is kept at 2 mph and the grade starts at 0 and inclines by 2% every two minutes.
Change in Ankle-Brachial Index (ABI) | Baseline, Month 3, Month 6, Month 9
  To obtain the ankle-brachial index (ABI), bilateral upper and lower extremity blood pressure cuffs are inflated about 30 millimeters of mercury (mmHg) above the systolic pressure. Doppler flow signals are used to detect the reappearing perfusion while reducing the cuff pressure. The results is expressed as a segmental/arm pressure ratio (ABI index). The highest pressure of the two arms will be used for calculating the ABI. The average ratio is about 1.0+/-0.10; an index of 0.90 or lower is considered abnormal. In patients with calcific, non-compressible arteries (certain diabetics) where ABI measurements are unreliable, a toe/ arm pressure index ratio will be performed, with a 2.5 cm cuff used on the great or second toes. A toe/arm index less than 0.65 is considered abnormal.
Change in Foot Transcutaneous Oxygen Tension (TcPO2) | Baseline, Month 3, Month 6, Month 9
  Foot transcutaneous oxygen tension (TcPO2) is a noninvasive way to measure peripheral arterial disease. TcPO2 is obtained with a monitor before exercise after the patients have been standing for three minutes and is monitored throughout exercise. Values are recorded at initial claudication distance, absolute claudication distance, and after recovery from exercise. A commonly used cut point is 60 millimeters of mercury (mmHg), with values below this indicating the presence of peripheral arterial disease.

CONTACTS AND LOCATIONS:
Overall Officials: Arshed Quyyumi, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta A, Mavromatis K, Ko YA, Rogers SC, Dhindsa DS, Goodwin C, Patel R, Martini MA, Prasad M, Mokhtari A, Hesaroieh IG, Frohwein SC, Kutner MH, Harzand A, Wells BJ, Duwayri Y, Alabi O, Rajani RR, Brewster LP, Waller EK, Quyyumi AA. Rationale and design of the granulocyte-macrophage colony stimulating factor in peripheral arterial disease (GPAD-3) study. Contemp Clin Trials. 2020 Apr;91:105975. doi: 10.1016/j.cct.2020.105975. Epub 2020 Mar 4. PMID 32145440